CLINICAL TRIAL: NCT03079583
Title: The Efficacy of Zinc-biofortified Rice in Improving Zinc Status in Young Bangladeshi Children, a Double Blind Randomized Controlled Trial
Brief Title: The Efficacy of Zinc-biofortified Rice in Bangladeshi Children
Acronym: ZARI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: HarvestPlus (Other); BRAC University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ZARI_1_trail
Record Dates: First submitted 2017-03-03; First posted 2017-03-14 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Zinc Deficiency; Growth; Stunting, Nutritional
Keywords: Zinc Biofortification; Zinc Status; Zinc Biomarker
MeSH Terms: conditions — Growth Disorders | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control-group (Placebo Comparator): Control Rice used for meal, normal zinc level
  Interventions: Dietary Supplement: Control-group
- Intervention-group (Active Comparator): Biofortified Rice used for meal, around 30% higher zinc level
  Interventions: Dietary Supplement: Intervention-group

INTERVENTIONS:
Dietary Supplement: Intervention-group — Biofortified Rice is grown by foliar Zn application
  Arms: Intervention-group
Dietary Supplement: Control-group — Control Rice with normal zinc levels
  Arms: Control-group

SUMMARY:
To assess the efficacy of the zinc biofortified rice on plasma zinc concentrations in infants from a rural area of Bangladesh.

DETAILED DESCRIPTION:
Rationale: Around the world and estimated 30% of the population is at risk of Zinc deficiency, mainly due to monotonous plant base diets and the poor bioavailability of this sources. One staple food crop which is low in zinc content is rice. Therefore, zinc deficiency is highly common in Asia. Zinc plays a major role in child growth and neurobehavioral development. Furthermore, it is linked to infection control and normal immune response. One way to add extra zinc to someone's diet is zinc bio fortification of staple crops, which can be a cost saving sustainable approach to improve zinc nutrition. However, data on long-term intake of biofortified crops with zinc is scarce and efficacy of newly developed rice crops high in zinc are not well known.

Objective: The objective is to assess the efficacy of a newly developed zinc biofortified rice variety on plasma zinc concentrations in children in a rural area of Bangladesh when compared to their controls in a 9 month randomized controlled trial (RCT).

Study design: A double randomized control trial. Study population: Stunted children whom are zinc deficient at start of the study intervention determined by plasma zinc levels <9.9 µmol/L.

Main study parameters/endpoints: The difference in zinc status between the intervention and control group expressed in blood plasma zinc levels. Plasma zinc will be measured 4 times during the intervention period. Besides plasma zinc other zinc biomarkers will be tested for their usefulness.

ELIGIBILITY:
Inclusion Criteria:

* 12-36 months of age (at baseline assessment)
* Low plasma Zn concentration (<10.71 µmol/L)
* Marginally stunted (height for age Z-score <-1.75)
* The informed consent form has been read and signed by the caregiver (or has been read out to the caregiver in case of illiteracy)

Exclusion Criteria:

* Severe Anemia (Hb< 70 g/L)
* Chronic or acute illness or other conditions that in the opinion of the Principle Investigator (PI) or co-researchers would affect Zn metabolism or would render the participant unable to comply with the protocol (based on self-reporting or diagnosed during screening)
* Participants taking part in other studies requiring the drawing of blood
* Not planning long-term residence in study site
* Regular intake (>2 days) of iron-containing mineral and vitamin supplements or fortified foods within the last 2 months
* Chronic use of drugs that affect the metabolism of Zn, including reducing absorption or increasing excretion; e.g., tuberculosis medications (ethambutal and isoniazides), drugs used as treatment for entamoeba hystolica (diiodohydroxyquin), drugs that reduce stomach acidity (H2 blockers and proton pump inhibitory), antidepressants (nialamide and socarboxazid), anti-inflammatory drugs (corticosteroids), diuretics (thiazides).

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 520 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2019-04-25 (Actual)

PRIMARY OUTCOMES:
plasma zinc | 4 collection points in total. 2 fixed at start and end of intervention (week 1&36, T=1,4). 2 sparse random sampling points (RSP) in-between T=1-4. First RSP between 2-5 months (week 5-20 T=2). Second RSP between 5-8 months (week 21-32,T=3).
  Change of plasma zinc values from baseline to endpoint and 2 times within study period

SECONDARY OUTCOMES:
Inflammatory markers | 4 collection points in total. 2 fixed at start and end of intervention (week 1&36, T=1,4). 2 sparse random sampling points (RSP) in-between T=1-4. First RSP between 2-5 months (week 5-20 T=2). Second RSP between 5-8 months (week 21-32,T=3).
  C reactive protein (CRP),alpha1-acid glycoprotein (AGP)
Length | 4 collection points in total. 2 fixed at start and end of intervention (week 1&36, T=1,4). 2 sparse random sampling points (RSP) in-between T=1-4. First RSP between 2-5 months (week 5-20 T=2). Second RSP between 5-8 months (week 21-32,T=3).
  Length (in cm) measurement for anthropometric (HAZ-scores).
Weight | 4 collection points in total. 2 fixed at start and end of intervention (week 1&36, T=1,4). 2 sparse random sampling points (RSP) in-between T=1-4. First RSP between 2-5 months (week 5-20 T=2). Second RSP between 5-8 months (week 21-32,T=3).
  Weight (in kg) measurement for anthropometric (HAZ-scores).
Morbidity | Fixed assessment once a week for every participant throughout the intervention period (week 1-36).
  diarrhea and disease episodes will be recorded weekly throughout the study
FADS analyses | Secondary analyses of collected plasma samples, in subset of participants (75 children from each group, random selected, matched baseline and endpoint samples)
  FADS plasma analyses for zinc biomarker determination
Iron status | 4 collection points in total. 2 fixed at start and end of intervention (week 1&36, T=1,4). 2 sparse random sampling points (RSP) in-between T=1-4. First RSP between 2-5 months (week 5-20 T=2). Second RSP between 5-8 months (week 21-32,T=3).
  Plasma ferritin
Iron status | 4 collection points in total. 2 fixed at start and end of intervention (week 1&36, T=1,4). 2 sparse random sampling points (RSP) in-between T=1-4. First RSP between 2-5 months (week 5-20 T=2). Second RSP between 5-8 months (week 21-32,T=3).
  Hemoglobin

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Zimmermann, Prof. Dr., Principal Investigator — Professor, Laboratory of Human Nutrition, Department of health science and technology, ETH Zurich, Zurich, Switzerland; Malay K Mridha, Assoc. Prof., Principal Investigator — Associate Professor, James P Grant school of Public Health, BRAC University, Dhaka, Bangladesh
Locations (2):
- BRACU, Bangladesh, Dhaka, Bangladesh
- Swiss Federal Institute of Technology (ETH), Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jongstra R, Hossain MM, Galetti V, Hall AG, Holt RR, Cercamondi CI, Rashid SF, Zimmermann MB, Mridha MK, Wegmueller R. The effect of zinc-biofortified rice on zinc status of Bangladeshi preschool children: a randomized, double-masked, household-based, controlled trial. Am J Clin Nutr. 2022 Mar 4;115(3):724-737. doi: 10.1093/ajcn/nqab379. PMID 34792094